CLINICAL TRIAL: NCT07035678
Title: A Study on the Associations of Toll-like Receptor 5 Gene Polymorphisms With Crohn's Disease in Chinese Patients
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2025-01-221
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Crohn's Disease; Ustekinumab; Toll-like Receptor 5; Polymorphism, Single Nucleotide
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Crohn's disease group: Diagnosed with Crohn's disease.
- Normal control group: Healthy individuals without a history of rheumatoid arthritis, systemic lupus erythematosus, intestinal tuberculosis, ischemic enteritis, radiation enteritis, tumors, etc.

SUMMARY:
The exact etiology and pathogenesis of Crohn's disease (CD) have not been fully elucidated, and may be related to the combined effects of genetics, environment, immunity, gut microbiota, and many other factors. Toll like receptor 5 (TLR5) is one of the transmembrane pattern recognition receptors that specifically recognizes and binds to bacterial flagellar proteins, activating the nuclear factor kappa-B (NF - κ B) signaling pathway and triggering immune and inflammatory responses. The TLR5 gene is located in the 1q33.3 region of the human chromosome, with a total length of approximately 34kb and 6 exons. Research data from European populations shows that two single nucleotide polymorphisms, rs5744168 and rs5744174, in the TLR5 gene may be closely associated with the risk of developing CD. According to Danish scholars, the mutation of rs5744174 may affect the clinical response of CD patients treated with anti-tumor necrosis factor - α (TNF - α) drugs.

Ustekinumab (UST) is a fully humanized monoclonal antibody against the p40 subunit and is one of the commonly used biologics for treating CD patients. The p40 subunit is a common component of interleukin-12 (IL) and IL-23, therefore UST can simultaneously inhibit the IL-12 and IL-23 signaling pathways, exerting anti-inflammatory effects by suppressing immune cell differentiation such as T helper cell 1 (Th1), Th17 cells, natural killer cells, macrophages, etc. Among CD patients receiving UST treatment, it was found that patients who achieved clinical response in the early stage were more likely to achieve clinical remission in the middle and later stages compared to those who did not , indicating that evaluating early response has certain clinical value in predicting the efficacy of UST in the middle and later stages. This study aims to explore the relationship between TLR5 (rs5744168 and rs5744174) gene polymorphism and the risk and clinical pathological characteristics of CD in the Han population of Zhejiang, and analyze whether TLR5 gene mutations affect the early response of UST treatment for CD patients. The aim is to provide some clues and basis for revealing the genetic and immunological pathogenesis of CD and developing precise individualized treatment plans for UST.

ELIGIBILITY:
Inclusion Criteria:

1. After receiving IFX conventional treatment plan for 30 weeks;
2. Not participated in any other experimental projects in the past three months;
3. There are no other serious and life-threatening diseases in various systems.

Exclusion Criteria:

1. Pregnancy;
2. Breastfeeding;
3. Severe drug allergy (having experienced severe drug allergic reactions such as anaphylactic shock, systemic dermatitis, etc.);
4. Merge with other autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, autoimmune thyroiditis);
5. Merge malignant tumors;
6. Serious cardiovascular and cerebrovascular diseases;
7. Poor patient compliance or presence of mental disorders;
8. Incomplete case data.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese
Sampling Method: Non-Probability Sample
Enrollment: 825 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Harvey Bradshaw Index | 8 weeks
  mild: 0 to 8, moderate: 9 to 16, severe: 17 to 25
TLR5 gene polymorphisms | 0 week

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China